CLINICAL TRIAL: NCT00256191
Title: A Phase 1, Open-Label, Q21 Day Dose Escalation, Multi-Center Study of TPI 287 in Patients With Advanced Malignancies
Brief Title: Study of TPI 287 Administered Every 21 Days in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortice Biosciences, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI 287-02
Expanded Access: Available
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2005-11

CONDITIONS: Neoplasms; Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: taxanes; multidrug resistance; mutant tubulin binding; Hodgkin's or Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TPI 287 Injection

SUMMARY:
Tapestry Pharmaceuticals, Inc. has developed a novel taxane analog, TPI 287. TPI 287 is synthetically manufactured from naturally occurring taxanes extracted from yew starting material. The synthesis involves modification to the taxane side chain to overcome multidrug resistance and to achieve mutant tubulin binding. This study will be a multi-center, dose escalation, sequential group, Phase 1 study evaluating the intravenous administration of TPI 287 on an every 21 day cycle.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the maximum tolerated dose of TPI 287 administered every 21 days for Phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Patients must be/have:

* Histological evidence of malignancy
* Advanced solid tumors that have recurred or progressed following standard therapy
* Failed one prior therapy or have no standard therapy available
* Ambulatory with ECOG of 0-1 and estimated life expectancy of > 3 months
* If female, negative pregnancy test
* If of childbearing years, agree to use birth control
* If patient with prior radiation therapy for brain metastases, on steroids, must have been stable for 1 month

Exclusion Criteria:

Patients will be excluded if they are or have had:

* Prior radiation within 4 weeks
* Active medical condition or organ disease which may compromise safety or interfere with the study
* Clinically significant cardiac co-morbidities or pulmonary impairment
* Concomitant therapy needs
* Treated with any investigational drugs within 30 days
* Tumors involve major artery or vein
* Prior or concurrent central nervous system (CNS) disease
* Less than 4 weeks since major surgery
* Known to be positive for HIV, hepatitis B or C
* Concurrent use of aspirin
* Use of thrombolytic agents
* Uncontrolled hypertension
* Grade II-IV peripheral vascular disease
* Pregnant or lactating
* Prior allergic history to compounds of similar chemical composition
* Inpatients
* Grade II-IV peripheral neuropathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of TPI 287 administered every 21 days

SECONDARY OUTCOMES:
To determine the safety of TPI 287
To determine the antitumor activity of TPI 287
To determine the pharmacokinetic profile of TPI 287

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, MD, Study Director — Tapestry Pharmaceuticals, Inc.
Locations (1):
- Rocky Mountain Cancer Center, Denver, Colorado, United States